CLINICAL TRIAL: NCT00892190
Title: A Phase 1, Open-label, Dose-escalation Study of Dasatinib and All-Trans Retinoic Acid for Relapsed/Refractory and/or Elderly Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Study of Dasatinib and All-Trans Retinoic Acid for Relapsed/Refractory and/or Elderly Patients With Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 08-160
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; Dasatinib; all trans retinoic acid; relapsed AML; refractory AML; Relapsed/Refractory Acute myelogenous leukemia; Elderly subjects (age 65 or older) with acute myelogenous leukemia; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Dasatinib; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dasatinib (SPRYCEL) and all trans retinoic acid (VESANOID) (Experimental): Dasatinib DL0 - 50 mg every 24 hours DL1 (START)- 70 mg every 24 hours DL2 - 100 mg every 24 hours DL3 - 140 mg every 24 hours
  ATRA 22.5mg/m2 every 12 hours
  Interventions: Drug: dasatinib (SPRYCEL); Drug: all trans retinoic acid (VESANOID)

INTERVENTIONS:
Drug: dasatinib (SPRYCEL) — DL0 - 50 mg every 24 hours DL1 (START)- 70 mg every 24 hours DL2 - 100 mg every 24 hours DL3 - 140 mg every 24 hours
Drug: all trans retinoic acid (VESANOID) — 22.5mg/m2 every 12 hours

SUMMARY:
This is an open label, prospective, single institution dose-escalation study. The patient population includes non-induction candidate elderly patients with AML or MDS and/or patients with high-risk or relapsed/refractory AML or MDS. Five dose cohorts will be evaluated using a fixed dose of ATRA in combination with an escalating dose of dasatinib. The investigators will treat with an escalating dose of dasatinib from 70mg to 140mg daily. Dose escalation will proceed in a standard 3+3 fashion. A de-escalation to a 50 mg total daily dose of dasatinib is planned if DLT is greater than or equal to 33% is observed at the first dose level. Once the MTD for the combination of the drugs has been established, up to 6 additional patients will be enrolled at the MTD level to obtain additional safety information about the combination and to allow for preliminary laboratory correlate analysis.

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the safety and tolerability of the combination of dasatinib and ATRA in relapsed or elderly, non-induction candidate acute myelogenous leukemia (AML) or MDS patients and to identify the maximally tolerated dose (MTD), dose-limiting toxicities (DLT).

Secondary Objectives:

1. To determine the pharmacokinetic (PK) profiles of dasatinib and ATRA when administered as combination therapy for patients with AML or MDS
2. To determine if the combination therapy of dasatinib and ATRA promotes differentiation of AML or MDS .

ELIGIBILITY:
Inclusion

* Informed consent
* Performance Status (ECOG) less than or equal to 3
* Subjects ages 18 or older
* Confirmed diagnosis of non-APL AML (WHO criteria) or high-risk MDS (IPSS criteria INT-2 or High)
* For subjects Age <65: Refractory AML or AML relapse within six months of attaining remission or AML relapse more than six months after achieving a remission, who cannot achieve a second remission or Untreated subjects who develop AML after preexisting hematologic disease or Secondary AML or high-risk MDS who either are not a candidate for hypomethylating agents or who have failed one or more hypomethylating agent
* For subjects Age ≥65: De novo AML not candidates for induction chemotherapy or Refractory AML or AML relapse within six months of attaining remission or AML relapse more than six months after achieving a remission, who cannot achieve a second remission or Untreated subjects who develop AML after preexisting hematologic disease Secondary AML or high-risk MDS who either are not a candidate for hypomethylating agents or who have failed one or more hypomethylating agent
* Life expectancy of at least 2 months
* Adequate Organ Function: Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN), Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN, Serum Creatinine < 2.0 times the institutional ULN
* Ability to take oral medication (dasatinib must be swallowed whole)
* Concomitant Medications: Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib). Patient agrees that IV bisphosphonates will be withheld for the 4 weeks of dasatinib therapy due to risk of hypocalcemia.
* Age and Sex: Men and women, age 18-100. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 30 days after the last dose of study drug to minimize the risk of pregnancy. WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as: Amenorrhea that has lasted for >= 12 consecutive months without another cause, or For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL. Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of the investigational product. A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study [and for up to 30 days after the last dose of study drug] to minimize the risk of pregnancy. A barrier method is recommended.

Exclusion:

* Sex and Reproductive Status: WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after the last dose of study drug. Women who are pregnant or breastfeeding. Women with a positive pregnancy test. Sexually active fertile men not using effective birth control if their partners are WOCBP.
* Target Disease Exceptions: Subjects with a diagnosis of Acute Promyelocytic Leukemia, Known or clinically suspected CNS involvement, HIV Positivity, A diagnosis of another active malignancy with the exception of non-melanoma skin cancer or cervical cancer in situ., Gastrointestinal conditions that could affect drug absorption including post surgical states such as gastric bypass, History of psychiatric disorder which may compromise compliance, Stem cell transplant within 60 days., Subjects who have undergone stem cell transplant who are undergoing treatment or prophylaxis for Graft versus host disease
* Medical History and Concurrent Diseases: Concurrent medical condition which may increase the risk of toxicity, including: Pleural or pericardial effusion of any grade, Cardiac Symptoms; any of the following will be considered for exclusion: Uncontrolled angina, congestive heart failure or MI within (6 months), Diagnosed congenital long QT syndrome, Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), Prolonged QTc interval on pre-entry electrocardiogram (> 470 msec), Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
* Physical and Laboratory Test Findings: Chronic diarrhea, Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
* Allergies and Adverse Drug Reactions: History of allergic reaction to ATRA, History of allergic reaction to dasatinib
* Prohibited Treatments and/or Therapies: Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes or prolonge QT interval including: (Patients must discontinue drug 7 days prior to starting dasatinib) (See section 5.6.1.2) quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine, azithromycin, citalopram, escitalopram, flecainide, mesoridazine, sevoflurane. Potent inhibitors of CYP3A4 (see section 5.6.1.1 for more details). Proton pump inhibitors and H2 inhibitors (see section 5.6.2.3). St. John's Wort (see section 5.6.2.4). Medications that inhibit platelet function and anticoagulants (see section 5.6.2.5). Currently receiving anticancer therapy. Use of hydroxyurea within 7 days prior to screening labs. Treatment with a an investigational agent within 30 days prior to the first dose of dasatinib/ATRA or planning to receive an investigational agent during the study. Growth factors within 14 days prior to screening labs
* Other Exclusion Criteria: Prisoners, or subjects who are involuntarily incarcerated. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and DLTs of dasatinib in combination with ATRA given the proposed dose escalation plan. | 1.5 years

SECONDARY OUTCOMES:
Assessment of Differentiation. Bone marrow biopsies and aspirates will be obtained pre-treatment, on day 14, and day 28. These will be subjected to morphologic, cytochemical, and routine flow cytometric analyses. | 1.5 years
Assess treatment effects on SFK (Src family kinase) activation and expression of RARA target genes. | 1.5 years
PK parameters including peak concentration (Cmax),Tmax, Cmin, the area under the curve (AUC), volume of distribution, clearance terms, elimination rate constant, and elimination half-life (t1/2) will be analyzed. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Redner, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Cancer Institute - Hillman Cancer Center, Pittsburgh, Pennsylvania, United States